CLINICAL TRIAL: NCT05502354
Title: A Single Arm Study to Investigate the Safety and Efficacy of C Reactive Protein (CRP) Guided Transanal Drainage Tube (TDT) Removal for Anastomotic Leak (AL) Prevention Following Laparoscopic Anterior Resection for Rectal Carcinoma
Brief Title: CRP-guided Transanal Drainage Removal After Rectal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, XIANG ZHANG, Principal Investigator, Qilu Hospital of Shandong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CRC-2022-01
Record Dates: First submitted 2022-08-11; First posted 2022-08-16 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Rectal Cancer; Anastomotic Leak
MeSH Terms: conditions — Rectal Neoplasms; Anastomotic Leak

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with TDT removal guided by postoperative CRP trajectory (Experimental)
  Interventions: Device: removal of transanal drainage tube

INTERVENTIONS:
Device: removal of transanal drainage tube — removal of transanal drainage tube after laparoscopic anterior resection for rectal carcinoma according to postoperative CRP trajectory

SUMMARY:
Transanal drainage tube (TDT) has the benefit of reducing intraluminal pressure after rectal surgery and may provide ideal regional environment for anastomotic healing. Postoperative C-reactive protein (CRP) trajectory has a high negative predictive value of 0.99 for ruling out anastomotic leak (AL). Previously, TDT was removed at the surgeon's own discretion. In the present study, we design a single arm study to investigate the safety and efficacy of CRP-guided TDT removal for AL prevention following laparoscopic anterior resection for rectal carcinoma

ELIGIBILITY:
Inclusion Criteria:

* age from 18 to 75 years old
* male and female
* primary rectal adenocarcinoma
* ASA I, II, or III
* laparoscopic LAR + DST
* with or without preoperative radio- or chemotherapy
* no distal metastasis
* no preoperative bowel obstruction
* no preventive ileostomy or colostomy
* patients and their families can understand and are willing to participate in this study and provide written informed consent

Exclusion Criteria:

* emergency operation
* preoperative abnormal liver function
* tatme or ISR procedure (healing process might differ from anterior resection)
* severe postoperative (Clavien-Dindo grade III IV V) complications other than anastomotic leak
* severe perioperative infection unrelated to anastomotic leak
* patients with serious mental illness
* pregnant or breastfeeding women
* patients with other clinical and laboratory conditions considered by the investigator should not participate in the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
anastomotic rate | 30 days after surgery
  anastomotic rate

SECONDARY OUTCOMES:
the grades of anastomotic leak | 30 days after surgery
  The severity grading of anastomotic leak according to the International Study Group of Rectal Cancer
rates of diarrhea after transanal drainage tube removal | from transanal drainage tube removal to 30 days after surgery
  rates of diarrhea after transanal drainage tube removal
visual analogue scale to assess anal postoperative pain | from the date of transanal drainage tube positioning until the tube is removed, assessed up to 2 weeks
  visual analogue scale of the included patients to assess the transanal drainage tube tolerability. Visual analogue scale ranges from 0-10. 0 indicates perfectly tolerated while 10 indicates complete intolerant and the tube has to be removed.
transanal drainage tube-related adverse events | from the date of transanal drainage tube positioning until the tube is removed, assessed up to 2 weeks
  transanal drainage tube-related adverse events such as bleeding and iatrogenic colonic perforations

CONTACTS AND LOCATIONS:
Overall Officials: Kexin Wang, M.D. Ph.D., Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided